CLINICAL TRIAL: NCT01836874
Title: Prophylaxis of Migraine Patients With Topiramate in India (PROMPT-IN)
Brief Title: A Study of Prophylaxis for Migraine Patients With Topiramate in India
Acronym: PROMPT-IN
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100585; TOPMATMIG4020 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2013-03-21; First posted 2013-04-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Migraine
Keywords: Migraine; Indian; Topiramate
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Topiramate
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Participants receiving topiramate 25 mg once-a-day for 1 week and later on, receiving increase dose up to 200 mg, twice-a-day, orally will be observed for 3 months.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of topiramate in preventing migraine among Indian participants requiring prophylaxis (measure taken to maintain health and prevent the spread of disease).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (study conducted at multiple sites) study. In this study approximately 209 participants will be observed. Participants receiving topiramate will be observed monthly for 3 months. Safety assessments will include evaluation of adverse events and body weight of the participants which will be monitored throughout the study. The total duration of this study will be approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants who experiencing migraine three or more times per month and require prophylaxis medication
* Participants having at least 6 months of migraine history (diagnosed as per international headache society criteria with or without aura)
* Other indications for migraine prophylaxis are: the use of acute treatment medication too frequently (more than 2 treatment days per week); an increasing frequency of headaches that are non-responsive to acute therapy; requiring rescue therapy more than once a month
* Participants who are seen to benefit from topiramate based upon the physician's judgment

Exclusion Criteria:

* Headaches other than migraine or episodic tension or sinus headaches or having headaches exceeding 15 days per month
* Onset of migraine after age 50
* An exclusively migraine aura without headache or a painful condition other than migraine pain
* Having significant history of unstable medical disease
* At risk in terms of the contraindication in the product insert of topiramate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Indian participants experiencing migraine
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 3 months
Number of adverse events | Up to 3 months
Number of participants with incidence of discontinuation of study medication | Up to 3 months
Reason for participant's discontinuation of study medication | Up to 3 months
Change from baseline in the body weight | Baseline (screening) to 3 months
Participant's overall assessment of topiramate at the end of the treatment period | Month 3
  Participant's overall assessment is assessed at the end of study on a 5-point scale wherein 1= Very Good, 2 = Good, 3 = No Change, 4 = Poor & 5 = Very Poor. Higher scores indicate worsening.
Physician's overall assessment of topiramate at the end of the treatment period | Month 3
  Physician's overall assessment is assessed at the end of study on a 5-point scale wherein 1= Very Good, 2 = Good, 3 = No Change, 4 = Poor & 5 = Very Poor. Higher scores indicate worsening.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.